CLINICAL TRIAL: NCT03616119
Title: The Prevalence of Gastroesophageal Reflux Disease in Azerbaijan
Brief Title: Gastroesophageal Reflux Disease in Azerbaijan
Status: Completed | Type: Observational
Sponsor: Sevda Aghayeva (Other)
Collaborators: Azerbaijan Medical University (Other)
Responsible Party: Sponsor-Investigator, Sevda Aghayeva, principal investigator, Azerbaijan Gastroenterology and Hepatology Association
Organization: Azerbaijan Gastroenterology and Hepatology Association (Other)
Other Study IDs: QastroHep
Record Dates: First submitted 2018-07-29; First posted 2018-08-06 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: gastoesophageal reflux disease; prevalence; Azerbaijan
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the prevalence of Gastroesophageal reflux disease in Azerbaijan. It is intended to evaluate the prevalence of the disease in the regions as well as the capital by cluster sampling ,ethitology and to compare the outcomes depending on the geographical location.

DETAILED DESCRIPTION:
It is an observational, nationwide study. The GERD questionnaire (1994) requested from Mayo clinic, was received and validated. The questionnaire was translated by 3 individuals from english to azeri and back trasnlated by 3 native english speakers.

Power analysis was performed. The research was presented for the approval to Ethical Committee of Azerbaijan Medical University.

Prior to the actual study, a pilot study with smaller number of participants was performed and the results were evaluated.

Cluster sampling methodology was provided by the statistical department of Azerbaijan Medical University.

110 employees were hired for using a survey in different regions of Azerbaijan. Written consent was obtained from every person evaluated. Statistical ananlysis was performed.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80
* Both genders
* Hearburn
* Belching
* Regurgitation

Exclusion Criteria:

* protom pomp inhibitor use
* antibiotic use in the last 4 weeks
* upper GI surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-80 age range
Study Population: Azerbaijan is divided by clusters with a definite numbers of individuals to take survey on reflux disease in the given age range and calculated by proportion of males and females.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of GERD in Azerbaijan | 1 year
  The prevalence of GERD in Azerbaijan was 22.7% with significant female predominance (26.1% vs 15.3%; p<0.0001). GERD was defined in 17 % for ages below 35; 22.7 % for 36-55 and 38.5 % for those who are above 56 that, accordingly, indicating that GERD becomes significant as age increases (p<0.0001). Reflux was observed in 18.1% of normal weight respondents (BMI 18.6-24.9), 25.6% of overweight (BMI 25-29.9), and in 30.4% of obese (BMI>30) individuals (p=0.001). Regarding marital status, the prevalence was the lowest in the single subjects' group (17%), close to average in the married group (23.8%), and the highest (41.7%) in divorced/widowed cases (p=0.003). Stress was significantly affecting GERD distribution, affecting 59.4% of all respondents (p<0.004).
GERD questionnaire (GERD) of Mayo case 1998- 019 | 1 year
  Observational study

CONTACTS AND LOCATIONS:
Overall Officials: Sevda Aghayeva, MD, Principal Investigator — Azerbaijan Gastroenterology and Hepatology Association
Locations (1):
- Azerbaijan Gastroenterology and hepatology Association, Baku, Nasimi, Azerbaijan